CLINICAL TRIAL: NCT06944379
Title: Phase 1, First-in-human, Double-blind, Placebo-controlled, Single Dose Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of ORKA-002 in Healthy Participants
Brief Title: ORKA-002-211 A Phase I Study to Evaluate ORKA-002 in Healthy Volunteers Following A Single Dose
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Oruka Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ORKA-002-211
Record Dates: First submitted 2025-04-15; First posted 2025-04-25 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteers
Keywords: ORKA-002; Phase 1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ORKA-002 (Experimental): Subcutaneous (SC) injection of ORKA-002
  Interventions: Drug: ORKA-002
- Placebo (Placebo Comparator): Subcutaneous (SC) injection of placebo comparator
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ORKA-002 — ORKA-002 is supplied as sterile solution to be administered by SC injection
  Arms: ORKA-002
Other: Placebo — Placebo solution to be administered at a matching volume by SC injection
  Arms: Placebo

SUMMARY:
This is a Phase 1, first-in-human study to evaluate the safety, tolerability, and pharmacokinetics of ORKA-002 in healthy participants.

DETAILED DESCRIPTION:
This is a single center, Phase 1, double-blind, placebo-controlled, randomized, first-in-human (FIH), single ascending dose study evaluating the safety, tolerability, pharmacokinetics (PK) of ORKA-002 in healthy volunteers. The study will enroll approximately 24 healthy volunteers. The ORKA-002 dose will be administered by a subcutaneous injection.

ELIGIBILITY:
Key Inclusion Criteria:

1. Healthy male or female participants
2. 18 to 65 years (inclusive) with a body mass index (BMI) 18 to 32 kg/m2 at Screening
3. Willing and able to remain at the study site unit for the duration of the confinement period and return for the outpatient visit(s)/s defined in the protocol
4. Using two methods of contraception (one being highly effective) from admission through the end of the study

Key Exclusion Criteria:

1. Any clinically significant medical condition or finding that, in the Investigator's opinion, is likely to unfavorably alter the risk of study participation, confound study results, or interfere with the study conduct or compliance.
2. Known history of illicit drug use or drug abuse or harmful alcohol use
3. Known history of frequent tobacco or vaping use within 2 years prior to screening
4. Unwilling to abstain from regular, continuous alcohol use or tobacco use as per protocol
5. History of severe allergic reactions or hypersensitivity
6. Actively nursing, lactating, pregnant, or plans to be pregnant
7. Use of any investigational drug therapy within 30 days prior to enrollment
8. Unable to comply with study requirements or in the opinion of the Investigator should not participate in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-emergent Adverse Events | Day 1 through 1 year
  Incidence of treatment-emergent adverse events and clinically significant changes from baseline in vital signs, electrocardiograms, and clinical laboratory parameters

SECONDARY OUTCOMES:
Maximum observed serum concentration of ORKA-002 | Day 1 through 1 year
  Cmax of ORKA-002
Time to Cmax (Tmax) of ORKA-002 | Day 1 through 1 year
  Tmax of ORKA-002
Area under the serum concentration-time curve (AUC) of ORKA-002 | Day 1 through 1 year
  Area under the curve from the time of dosing to infinity (AUC0-inf)
Terminal elimination half-life (T1/2) | Day 1 through 1 year
  T1/2 of ORKA-002

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Breitschwerdt, Study Director — Oruka Therapeutics, Inc.; Principal Investigator, Principal Investigator — Oruka Therapeutics Investigative Site
Locations (1):
- Oruka Therapeutics Investigative Site, Christchurch, New Zealand, New Zealand